CLINICAL TRIAL: NCT04058600
Title: Exposure to Virtual Reality as Psychosocial Intervention in Colorectal Cancer Surgery in Hospital Clinic of Barcelona, Spain
Brief Title: Exposure to Virtual Reality as Psychosocial Intervention in Colorectal Cancer Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Antonio M Lacy, Chief of Gastrointestinal Surgery Department, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HCB/2018/0290 CIF-G-08431173
Record Dates: First submitted 2019-06-07; First posted 2019-08-15 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Anxiety; Colorectal Cancer
Keywords: virtual reality (VR); anxiety; colorectal cancer; surgery
MeSH Terms: conditions — Anxiety Disorders; Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Single center prospective randomized two arms study
Masking Description: No masking.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality (Experimental): The patients will be exposed to a virtual reality software that simulates the environment of the hospital, from admission to the operating room and the recovery room.
  Interventions: Behavioral: Virtual Reality Software
- Control (No Intervention): Patients in this group are not exposed preoperatively to the virtual reality software and are given the standard therapy and cares for their disease.

INTERVENTIONS:
Behavioral: Virtual Reality Software — Patients will be exposed to a virtual reality software that simulates the hospital environment, from admission to the operating room and the recovery room.
  Arms: Virtual Reality

SUMMARY:
A prospective controlled randomized interventional study comparing the effects of the preoperative exposure to a virtual reality software versus not exposure in 126 patients with colorectal cancer. Patients will be divided in two randomized groups, each of them of 63 patients. The hypothesis of the study is that gradual exposure to the hospital environment using a virtual reality software is effective to reduce preoperative anxiety.

The main variable is the level of anxiety in patients undergoing colorectal cancer surgery. It will be measured using State-Trait Anxiety Inventory Scale (STAI-S) and the Hospital Anxiety and Depression Scale (HADS).

DETAILED DESCRIPTION:
Colorectal cancer is the third most frequent neoplasia diagnosed worldwide, and in Spain it is the first in incidence and prevalence, accounting for 15% of all neoplasias according to World Health Organization (WHO).

The incidence of preoperative anxiety in patients undergoing elective surgery is high (60% - 76%). There are many causes for this: anticipation of postoperative pain, loss of independence, separation from the family, fear to the surgical procedure or to severe complications or even death. The incidence of preoperative anxiety varies according to age, sex, educational leve, previous exposure to surgical interventions and the expected impact of the surgical procedure in global quality of life.

Patients with anxiety require higher dosis of induction anesthesia, longer hospital stay, and a higher rate of perioperative complications due to a release of catecholamines, increase on the oxidative demands, causing tachycardia, arrhythmia, high blood pressure, etc.

Gradual exposition is considered an effective way of reducing anxiety. It has been demonstrated that anxiety is decreased in patients with history of surgical interventions, and thus the experience is experimented as an adaptive process. Virtual reality gives the opportunity to experience each of the steps of the hospital stay in a realistic environment.

The hypothesis of this study is that gradual exposure to the hospital environment using virtual reality is an effective tool to reduce preoperative anxiety in patients undergoing colorectal cancer surgery.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed of colorectal cancer requiring elective surgery.
* American Society of Anesthesiologists (ASA) I - III.
* No surgical history.
* Surgical procedure programmed in the next 6 months.

Exclusion Criteria:

* Neurologic deficits.
* Visual disorder.
* Neuro-psychiatric disorder.
* Use of neuro-psychiatric drugs.
* Non-sphincter-preserving surgery.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2018-04-11 (Actual); Primary Completion 2020-02-11 (Actual); Study Completion 2020-02-12 (Actual)

PRIMARY OUTCOMES:
State-Trait Anxiety Inventory (STAI) | 1 day prior to surgical intervention
  Change from Baseline Anxiety STAI scale to STAI scale the day previous to the surgery. Range of scores for each subtest is 20-80, the higher score indicating greater anxiety.
Hospital Anxiety and Depression Scale (HAD) | 1 day prior to surgical intervention
  Change from Baseline Anxiety HAD to HAD scale the day previous to the surgery. The total score for the HADS-A can range from 0 to 21. The following guidelines are recommended for the interpretation of scores: 0-7 for normal or no anxiety, 8-10 for mild anxiety, 11-14 for moderate anxiety, and 12-21 for severe anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- Victor Turrado-Rodriguez, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) data will not be available to other researchers. The study protocol and the global data will be available in the written paper.

REFERENCES:
- [Background] Romanik W, Kanski A, Soluch P, Szymanska O. [Preoperative anxiety assessed by questionnaires and patient declarations]. Anestezjol Intens Ter. 2009 Apr-Jun;41(2):94-9. Polish. PMID 19697827
- [Background] Matthias AT, Samarasekera DN. Preoperative anxiety in surgical patients - experience of a single unit. Acta Anaesthesiol Taiwan. 2012 Mar;50(1):3-6. doi: 10.1016/j.aat.2012.02.004. Epub 2012 Mar 30. PMID 22500906
- [Background] Tulgar S, Boga I, Piroglu MD, Ates NG, Bombaci E, Can T, Selvi O, Tas Z, Kose HC. Preoperative Anxiety before Spinal Anesthesia: Does Internet-based Visual Information/Multimedia Research Decrease Anxiety and Information Desire? A Prospective Multicentered Study. Anesth Essays Res. 2017 Apr-Jun;11(2):390-396. doi: 10.4103/0259-1162.206278. PMID 28663628
- [Background] Marcolino JA, Suzuki FM, Alli LA, Gozzani JL, Mathias LA. [Measurement of anxiety and depression in preoperative patients. Comparative study.]. Rev Bras Anestesiol. 2007 Apr;57(2):157-66. doi: 10.1590/s0034-70942007000200004. Portuguese. PMID 19466349
- [Background] Jafar MF, Khan FA. Frequency of preoperative anxiety in Pakistani surgical patients. J Pak Med Assoc. 2009 Jun;59(6):359-63. PMID 19534368
- [Background] Santos LJ, Garcia JB, Pacheco JS, Vieira EB, Santos AM. Quality of life, pain, anxiety and depression in patients surgically treated with cancer of rectum. Arq Bras Cir Dig. 2014 Apr-Jun;27(2):96-100. doi: 10.1590/s0102-67202014000200003. PMID 25004285
- [Background] Kaur H, Singh G, Singh A, Sharda G, Aggarwal S. Evolving with modern technology: Impact of incorporating audiovisual aids in preanesthetic checkup clinics on patient education and anxiety. Anesth Essays Res. 2016 Sep-Dec;10(3):502-507. doi: 10.4103/0259-1162.177187. PMID 27746541
- [Background] Eijlers R, Legerstee JS, Dierckx B, Staals LM, Berghmans J, van der Schroeff MP, Wijnen RM, Utens EM. Development of a Virtual Reality Exposure Tool as Psychological Preparation for Elective Pediatric Day Care Surgery: Methodological Approach for a Randomized Controlled Trial. JMIR Res Protoc. 2017 Sep 11;6(9):e174. doi: 10.2196/resprot.7617. PMID 28893727
- [Background] Ortuno-Sierra J, Garcia-Velasco L, Inchausti F, Debbane M, Fonseca-Pedrero E. New approaches on the study of the psychometric properties of the STAI. Actas Esp Psiquiatr. 2016 May;44(3):83-92. Epub 2016 May 1. PMID 27254400